CLINICAL TRIAL: NCT00683163
Title: PTH & Ibandronate Combination Study (PICS): Optimizing the Use of PTH With Boniva (Pilot Randomized Controlled Trial)
Brief Title: PTH & Ibandronate Combination Study (PICS)
Acronym: PICS
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PICS001
Record Dates: First submitted 2008-05-20; First posted 2008-05-23 (Estimated); Results first posted 2013-11-05 (Estimated); Last update posted 2013-11-05 (Estimated); Status verified 2013-08

CONDITIONS: Osteoporosis
Keywords: Combination of PTH and ibandronate; Bone marker formation; Postmenopausal; Trabecular spine BMD
MeSH Terms: conditions — Osteoporosis | interventions — Parathyroid Hormone; Ibandronic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A: 6 months both + 18 months oral only (Active Comparator): Group A will receive 6 months of monthly oral ibandronate 150 mg, plus daily PTH 1-84, 1.4 mg; followed by 18 months of ibandronate only. Placebo injections will be given months 13-15. Calcium + Vitamin D supplements, plus multivitamins are provided.
  Interventions: Drug: PTH(1-84); Drug: Ibandronate; Other: Placebo injection
- B: (3 months injection + 9 months oral) x 2 years (Active Comparator): Group B will receive 3 months of daily PTH 1-84, 1.4 mg; followed by 9 months of monthly oral ibandronate, 150 mg in year 1. In year 2, the group will receive another 3 months of daily PTH 1-84; followed by 9 months of monthly ibandronate. Placebo monthly pills will be given months 1-3 and months 13-15, and placebo injections will be given months 4-6. Calcium + Vitamin D supplements, plus multivitamins are provided.
  Interventions: Drug: PTH(1-84); Drug: Ibandronate; Other: Placebo injection; Other: Placebo pills

INTERVENTIONS:
Drug: PTH(1-84) — 1.4 mg injected subcutaneously (in the abdomen) daily
  Other Names: In Europe, PTH(1-84) is marketed as Preotact.
Drug: Ibandronate — 150mg by mouth once monthly
  Other Names: Boniva
Other: Placebo injection — Daily injections as placebo for PTS 1-84
Other: Placebo pills — Monthly pills as placebo for oral ibandronate
  Arms: B: (3 months injection + 9 months oral) x 2 years

SUMMARY:
This study will test in several innovative ways, several different combinations of PTH and oral monthly ibandronate for the treatment of osteoporosis in postmenopausal women. The intension is to provide other options for treatment than the current standard 2 year course of drug therapy. These options may lead to treatment where the two years of therapy are spread over several years.

DETAILED DESCRIPTION:
This randomized double-blind clinical trial for the treatment of postmenopausal osteoporosis will be conducted and coordinated by study investigators who also participated in the investigator-initiated PaTH study. Final data analysis will compare the results from this trial with those from the PaTH study. In the PaTH study, 238 women between 55 and 85 years of age were randomized to receive either:

1. PTH for 1 year followed by alendronate for 1 year
2. PTH and alendronate for 1 year followed by alendronate for 1 year
3. alendronate for 2 years
4. PTH for 1 year followed by placebo for 1 year.

In the PICS 44 postmenopausal women between the ages of 55 to 75 years of age with osteoporosis who meet the inclusion/exclusion criteria,will be randomized to the following 2 treatment groups. Group A will received 6 months of monthly Ibandronate, plus daily PTH 1-84,100 μg; followed by 18 months of Ibandronate only. Group B will received 3 months of daily PTH 1-84,100 μg; followed by 9 months of monthly Ibandronate, over 2 years. Calcium (400-650 mg) and Vitamin D (400 IU) supplements will be provided to all participants.

The primary objective is to determine if, at 3 months, the women treated with the concurrent combination of PTH and ibandronate (Group A) show a significant increase in bone marker formation compared to baseline (unlike the combination PTH/alendronate-treated women in PaTH). This will be accessed by examining the change in the markers P1NP, BSAP and serum CTX.

As a secondary objective, we will compare the trabecular spine BMD measures of those treated with concurrent PTH/Ibandronate (Group A) to those who received 3 months of PTH followed by Ibandronate(Group B). Another secondary objective will be to compare changes between groups in trabecular bone and DXA spine BMD after 2 years of treatment.

Changes to the fat content of the vertebrae during a course of PTH therapy will be examined using MRI spinal spectroscopy. Crosstabulation of these changes against changes in trabecular BMD, should indicate an effect on measurements. As well, the effect of a second three-month course of PTH therapy in Group B is of major interest.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Aged 55-75 years, inclusive, at randomization
* Postmenopausal for >= 5 years (no menses for at least 5 years)
* Have an evaluable bone mineral density scan (DXA) at the spine AND at the hip with a T-score <= -1.5 either at the spine or the femoral neck or total hip OR have a T-score <= -1.0 with at least one of the following risk factors for fracture: 1)Age >= 65 years; 2)History of post-menopausal fracture (non-vertebral or vertebral); 3)Maternal history of hip fracture.
* Be willing and able to self-administer daily injections
* Signed written consent form.

Exclusion Criteria:

* History of more than 12 months of oral bisphosphonate use ever, or any use (>4 weeks) with the past 12 months. For those with 4 weeks to 12 months of previous use, a 24 month washout is required.
* History of any IV bisphosphonate use.
* History of more than 12 month of PTH use ever, or any use (>4 weeks) with the past 12 months.
* History of estrogen (oral or patch) more than one month in the last 6 months or for more than 12 months in the last 2 years.
* Have type 1 or uncontrolled type 2 diabetes mellitus (defined as hemoglobin A1C > 10.0), or currently using insulin.
* Have serum calcium >10.2 mg/dl.
* Have Vitamin D level <15 nanograms/ml.
* Have Stage III renal insufficiency where calculated creatinine clearance < 40 ml/min by MDRD.
* Have any history of kidney stones in the last 10 years.
* Have any history of hypercalcuria or currently have urine calcium >300 mg/24 hours.
* Have any history of hypercalcemia.
* Have any history of sarcoidosis.
* Have any history of hyperparathyroidism.
* Have any history of active or treated tuberculosis or other granulomatous disorders.
* History of breast cancer, melanoma or hematologic malignancy which has required treatment within the last 10 years.
* Any history of bone cancer or Paget's disease of bone
* Any other metabolic bone disease which has required treatment within the last 10 years.
* History of any other non-skin cancer which has required treatment within the last 10 years.
* Have a documented history of symptomatic esophageal reflux, achalasia or esophageal stricture.
* Be currently taking > 7.5 mg systemic prednisone or equivalent per day or for more than 10 days in the last 3 months.
* Be currently using > 2 puffs, 4 times / day of inhaled steroids.
* Be currently taking anticoagulants.
* Be currently taking anticonvulsants that alter hepatic vitamin D clearance
* Have used Calcitonin within the past 3 months.
* Have used Raloxifene in the last 6 months or for more than 12 months in the last 2 years.
* Have used Tamoxifen in the last 6 months or for more than 12 months in the last 2 years.
* Have used fluoride for at least a month within the past 5 years.
* Be currently taking > 1000 IU/day Vitamin D
* Using Vitamin D analogues or metabolites.
* Be currently taking thyroid hormone replacement AND have a TSH < 0.1mIU/L.
* Have any major life-threatening illness.
* Concurrent enrollment in another double-blinded clinical treatment intervention study.
* Life expectancy less than 3 years
* Willing to discontinue all over the counter nutritional supplements

Ages: 55 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2008-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dennis M. Black, PhD, Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

REFERENCES:
- [Background] Li X, Kuo D, Schafer AL, Porzig A, Link TM, Black D, Schwartz AV. Quantification of vertebral bone marrow fat content using 3 Tesla MR spectroscopy: reproducibility, vertebral variation, and applications in osteoporosis. J Magn Reson Imaging. 2011 Apr;33(4):974-9. doi: 10.1002/jmri.22489. PMID 21448966
- [Result] Schafer AL, Burghardt AJ, Sellmeyer DE, Palermo L, Shoback DM, Majumdar S, Black DM. Postmenopausal women treated with combination parathyroid hormone (1-84) and ibandronate demonstrate different microstructural changes at the radius vs. tibia: the PTH and Ibandronate Combination Study (PICS). Osteoporos Int. 2013 Oct;24(10):2591-601. doi: 10.1007/s00198-013-2349-y. Epub 2013 Apr 16. PMID 23589163
- [Result] Schafer AL, Sellmeyer DE, Palermo L, Hietpas J, Eastell R, Shoback DM, Black DM. Six months of parathyroid Hormone (1-84) administered concurrently versus sequentially with monthly ibandronate over two years: the PTH and ibandronate combination study (PICS) randomized trial. J Clin Endocrinol Metab. 2012 Oct;97(10):3522-9. doi: 10.1210/jc.2012-1844. Epub 2012 Jul 12. PMID 22791766

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment letters were sent to women in the San Francisco Bay Area. Telephone screening interviews were conducted and study visits were performed at the San Francisco UCSF's Mt. Zion Medical Center.
Pre-assignment Details: Approximately 33,000 recruitment letters were mailed to women in the San Francisco Bay Area. Approximately 1100 phone calls were fielded, and 226 women were interested and eligible for additional screening. Of 164 who attended screening visits, 44 were eligible and enrolled.
Groups:
- Concurrent (A): Concurrent Group (A) received 6 months of monthly oral ibandronate 150 mg plus daily parathyroid hormone (PTH) 1-84 1.4 mg, followed by 18 months of ibandronate only. Placebo injections were given months 13-15.
- Sequential (B): Sequential Group (B) received 3 months of daily PTH 1-84 1.4 mg followed by 9 months of monthly oral ibandronate 150 mg in each of years 1 and 2. Placebo monthly pills were given months 1-3 and months 13-15, and placebo injections were given months 4-6.
Period: Overall Study
Arm/Group | Concurrent (A) | Sequential (B)
Started | 22 | 22
Completed | 22 | 22
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Concurrent (A): Concurrent Group (A) received 6 months of monthly oral ibandronate 150 mg plus daily PTH 1-84 1.4 mg, followed by 18 months of ibandronate only. Placebo injections were given months 13-15.
- Total: Total of all reporting groups
Arm/Group | Concurrent (A) | Sequential (B) | Total
Number analyzed (Participants) | 22 | 22 | 44
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 14 | 18 | 32
  >=65 years | 8 | 4 | 12
Age Continuous [Mean (Standard Deviation); unit: years] | 62.7 (4.1) | 61.2 (4.1) | 61.9 (4.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 22 | 44
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 22 | 22 | 44

OUTCOME MEASURES:

1. Primary Outcome: P1NP (ng/ml) Change From Baseline.
Description: After an overnight fast, serum was drawn at baseline and 1, 3, 6, 12, 15, 18 and 24 months. Samples were stored at -70C until batch assayed in a central laboratory. Serum N-propeptide of type I collagen (P1NP) and C-terminal telopeptide of type I collagen (CTX) were measured by electrochemiluminescent immunoassay. Bone-specified alkaline phosphate (BAP) was measured by paramagnetic particle immunoassay. P1NP was the bone turnover marker upon which we based sample size calculations.
Time Frame: Baseline, 3 months
Population: Analyses were performed according to intention-to-treat principle. A sample size of 20 participants per group was estimated to provide 80% power to detect a change of 25ng/mL in PINP, assuming the SD of 40ng/mL observed previously with concurrent PTH(1-84) and daily alendronate.
Measure: Geometric Mean (95% Confidence Interval); unit: Percent change from baseline
Groups:
- Concurrent (A): The Concurrent Group (A) received 6 months of monthly oral ibandronate 150 mg plus daily PTH 1-84 1.4 mg, followed by 18 months of ibandronate only. Placebo injections were given months 13-15.
- Sequential (B): The Sequential Group (B) received 3 months of daily PTH 1-84 1.4 mg, followed by 9 months of monthly oral ibandronate 150 mg in year 1 and again in year 2. Placebo monthly pills were given months 1-3 and months 13-15, and placebo injections were given months 4-6.
Arm/Group | Concurrent (A) | Sequential (B)
Number analyzed (Participants) | 22 | 22
Percent change from baseline | 42 [9 to 85] | 186 [119 to 275]

2. Secondary Outcome: Change From Baseline in Trabecular Spine vBMD
Description: Areal bone mineral density (aBMD) at the lumbar spine, hip, and distal one-third radius was assessed by dual-energy X-ray absorption at baseline and 6, 12, 18, and 24 months. The precision for aBMD is 1.0%. Volumetric BMD and bone geometry in trabecular and cortical compartments were assessed by quantitative computed tomography (QCT) at the spine and hip. The left hip was used for analysis. The precision for trabecular spine vBMD measurement is 1.0%. Trabecular spine vBMD was our primary BMD outcome, thus the one presented here.
Time Frame: Baseline, 24 months.
Measure: Mean (Standard Deviation); unit: Percent change from baseline
Arm/Group | Concurrent (A) | Sequential (B)
Number analyzed (Participants) | 22 | 22
Percent change from baseline | 12.5 (11.2) [119 to 275] | 13.7 (21.1) [138 to 300]
Statistical Analysis 1: Comparison: Concurrent (A) vs Sequential (B); Mean difference in percent change from baseline (Concurrent - Sequential); Test type: Superiority or Other; p = 0.82, t-test, 2 sided; Mean Difference (Net) = -1.2, 95% CI 2-sided [-11.5 to 9.2]

ADVERSE EVENTS:
Time Frame: Adverse event data was collected for the duration of the study (2 years) for each participant.
Arm/Group | Concurrent (A) | Sequential (B)
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 21/22 | 21/22
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Concurrent (A) (N=22) | Sequential (B) (N=22)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 5
Dizziness (General disorders) | 2 | 3
Fatigue (General disorders) | 3 | 1
Headache (General disorders) | 1 | 2
Limb Pain (Musculoskeletal and connective tissue disorders) | 5 | 6
Myalgia (General disorders) | 2 | 4
Abdominal Discomfort (Gastrointestinal disorders) | 4 | 1
Esophageal Reflux (Gastrointestinal disorders) | 2 | 3
Lower GI (Gastrointestinal disorders) | 5 | 5
Upper GI, Nausea/Vomiting (Gastrointestinal disorders) | 7 | 7
Upper GI, Other (Gastrointestinal disorders) | 2 | 3
Labs of Interest, Hypercalcemia (Blood and lymphatic system disorders) | 4 | 3
Labs of Interest, Hypercalciuria (Blood and lymphatic system disorders) | 2 | 1
Allergy (General disorders) | 2 | 1
Genitourinary (Renal and urinary disorders) | 1 | 3
Other (General disorders) | 7 | 6
Injection Site Complication (Injury, poisoning and procedural complications) | 6 | 8
Fracture (Injury, poisoning and procedural complications) | 1 | 3
Infection, Other (Infections and infestations) | 2 | 0
Infection, Upper Respiratory (Infections and infestations) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No